CLINICAL TRIAL: NCT01755247
Title: A Phase One, Single-Center, Open-Label, Randomized, Parallel Group, 3 Day Study Evaluating the Safety and Cutaneous Tolerability of NVN10000 Topical Gel in Healthy Volunteers
Brief Title: A Phase 1, 3 Day Study of Safety and Tolerability of NVN1000 Topical Gel in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NI-AC004
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-05

CONDITIONS: Acne Vulgaris
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Gels; berdazimer sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Topical Gel Vehicle (Placebo Comparator): Once daily application of topical gel vehicle to forehead for 3 days
  Interventions: Drug: Topical Gel Vehicle
- 8% NVN1000 Topical Gel (Active Comparator): Once daily application of 8% NVN1000 Topical Gel to the forehead for 3 days
  Interventions: Drug: 8% NVN1000 Topical Gel
- 8% NVN1000 Topical Gel and moisturizer (Active Comparator): Once daily application of 8% NVN1000 Topical Gel to the forehead, followed 15 minutes later by application of a commercially available moisturizer
  Interventions: Drug: 8% NVN1000 Topical Gel and moisturizer

INTERVENTIONS:
Drug: Topical Gel Vehicle
  Other Names: Vehicle
  Arms: Topical Gel Vehicle
Drug: 8% NVN1000 Topical Gel
  Other Names: NVN1000 Topical Gel
  Arms: 8% NVN1000 Topical Gel
Drug: 8% NVN1000 Topical Gel and moisturizer
  Other Names: NVN1000 plus moisturizer
  Arms: 8% NVN1000 Topical Gel and moisturizer

SUMMARY:
A Phase I, Single-Center, Open-Label, Randomized, Parallel Group, 3 Day Study Evaluating the Safety and Cutaneous Tolerability of NVN1000 Topical Gel in Healthy Volunteers

DETAILED DESCRIPTION:
This is a 3 day study to assess safety and tolerability of a new topical gel product, NVN1000 with and without the application of a commercially available moisturizer in approximately 15 healthy subjects. The test product will be applied to the forehead of healthy volunteers once daily for 3 days. One group of subjects will have a moisturizer applied to the same area 15 minutes after the test gel was applied and one group of subjects will be treated with the gel vehicle which does not contain the active product. The hypothesis is that the application of moisturizer will not effect safety or local tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male and Females > 18 years of age
* High degree of fluorescence of facial skin under Wood's lamp

Exclusion Criteria:

* Acute or chronic skin disorders
* Topical or systemic antibiotics within 4 weeks of study enrollment
* Use of medication that increases risk of methemoglobinemia or influences P. acnes counts
* Subjects with medical illnesses, anemia, elevated methemoglobin
* Women who are pregnant, nursing or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cutaneous tolerability | 3 days
  Tolerability based on a four point scale (0-3) for erythema, scaling ,dryness, pruritus, and burning/stinging.

SECONDARY OUTCOMES:
Safety comparison | 3 Days
  Assess safety through the comparison of adverse events between groups (lab assessments, physical exams and vital signs).

OTHER OUTCOMES:
Propionibacterium acnes counts | 3 days
  P. acnes counts will be obtained at Baseline, Day 1, and Day 3. The change in P acnes counts over time by treatment group will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: James J Leyden, Principal Investigator — KGL, Inc.
Locations (1):
- KGL, Inc, Broomall, Pennsylvania, United States